CLINICAL TRIAL: NCT03923023
Title: Preterm Resources, Education, and Effective Management for Infants
Brief Title: Impact of the PREEMI Package on Neonatal Mortality
Acronym: PREEMI
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Centre for Infectious Disease Research in Zambia (Other)
Responsible Party: Principal Investigator, Albert Manasyan, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: 14-F0023
Record Dates: First submitted 2019-04-15; First posted 2019-04-22 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Preterm Birth; Preterm Labor; Neonatal Death
Keywords: Facility delivery; Neonatal mortality; Preterm delivery; Preterm birth; Perinatal mortality
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature; Perinatal Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 42 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this Quality Improvement initiative is to reduce severe morbidity and mortality among premature infants through proven and cost-effective clinical management during the antenatal, intrapartum, and postpartum periods. In order to reduce neonatal mortality and morbidity due to preterm birth complications, health facilities must be able to identify and manage women in preterm labor, accurately administer medications, and provide high-quality postnatal care.

DETAILED DESCRIPTION:
The purpose of this Quality Improvement initiative is to reduce severe morbidity and mortality among premature infants through proven and cost-effective clinical management during the antenatal, intrapartum, and postpartum periods. In order to reduce neonatal mortality and morbidity due to preterm birth complications, health facilities must be able to identify and manage women in preterm labor, accurately administer medications, and provide high-quality postnatal care.

The study will provide evidence of implementing a package of clinical interventions coupled with quality improvement and monitoring strategy aimed at reducing neonatal mortality in 3 resource-limited health facilities, leveraging on an existing strengthened birth registry to provide neonatal outcomes up to 28 days after delivery. Additionally, using a multifaceted approach through an interdisciplinary team, the investigators will identify the social and cultural barriers that contribute to home-based deliveries. These findings will be helpful to the Ministry of Health in shaping future policies regarding the scale-up of newborn care clinical protocols as part of Government's efforts to reducing neonatal mortality in Zambia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who seek Antenatal care services and plan to deliver in the selected health facilities
* Women who reside within the larger catchment area of the selected 3 health facilities

Exclusion Criteria:

* Women who reside outside the larger catchment area of the health facilities
* Women who have not sought antenatal care services in the 3 health facilities and have come to only deliver there

Min Age: 10 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women who seek antenatal care and delivery services at the selected 3 health facilities.
Study Population: Pregnant women who seek antenatal care and delivery services at the selected 3 health facilities.
Sampling Method: Non-Probability Sample
Enrollment: 11195 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
10% relative risk reduction in 28-day neonatal mortality rate in preterm infants | Baseline to 36 months
  Rate of 28-day neonatal mortality at the end of the study compared to that at baseline

SECONDARY OUTCOMES:
20% relative risk reduction in all-cause 7-day neonatal mortality in preterm infants | Baseline to 36 months
  Rate of 7-day neonatal mortality at the end of the study compared to that at baseline
Factors that contribute to home and facility deliveries within the PREEMI facility catchment areas through the use of pre-determined questionnaire. | Baseline to 36 months
  Number of study participants who delivered at home and at a health facility

CONTACTS AND LOCATIONS:
Overall Officials: Albert Manasyan, MD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- Zambia (2):
  - Chawama 1st Level Hospital, Chipata 1st Level Hospital, and George Clinic, Lusaka
  - University Teaching Hospital, Lusaka

IPD SHARING:
Plan to Share IPD: Yes
The study data will be shared upon a reasonable request to the study PI.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be shared with the requesting investigator/entity.
Access Criteria: For secondary analysis purposes or verification of publication results.

REFERENCES:
- [Derived] Muttau N, Mwendafilumba M, Lewis B, Kasprzyk K, Travers C, Menon JA, Mutesu-Kapembwa K, Mangangu A, Kapesa H, Manasyan A. Strengthening Kangaroo Mother Care at a tertiary level hospital in Zambia: A prospective descriptive study. PLoS One. 2022 Sep 1;17(9):e0272444. doi: 10.1371/journal.pone.0272444. eCollection 2022. PMID 36048848
- [Derived] Tembo T, Koyuncu A, Zhuo H, Mwendafilumba M, Manasyan A. The association of maternal age with adverse neonatal outcomes in Lusaka, Zambia: a prospective cohort study. BMC Pregnancy Childbirth. 2020 Nov 11;20(1):684. doi: 10.1186/s12884-020-03361-5. PMID 33176718